CLINICAL TRIAL: NCT04278716
Title: Safe Return to Play Following Surgery for Labral Repair: Development and Validation of a Return to Play Checklist
Brief Title: Return to Play Checklist
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Rothman Institute Orthopaedics (Other)
Responsible Party: Sponsor
Other Study IDs: 2020 TJ 04
Record Dates: First submitted 2020-02-18; First posted 2020-02-20 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Labral Tear, Glenoid
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Utilization of a safe return to play checklist: Athletes who were treated for a capsulolabral tear who have undergone arthroscopic capsulolabral repair surgery will be evaluated using an objective checklist prior to being allowed to return to their sport. The utilization and outcome of using this checklist will be evaluated
  Interventions: Other: Safe return to play checklist

INTERVENTIONS:
Other: Safe return to play checklist — this objective checklist will be utilized by the physical therapy staff and surgeon to determine whether an athlete is safe to return to their sport

SUMMARY:
This study will try to develop and determine objective and validated criteria for our athletes to safely return to sports after labral repair.

ELIGIBILITY:
Inclusion Criteria:

- Males and non-pregnant females aged 15 years or older with a capsulolabral tear undergoing arthroscopic capsulolabral repair surgery at the Rothman Institute with one of the investigators

Exclusion Criteria:

* Patients with an labral repair
* Patients only undergoing debridements with no repair
* Patients undergoing revision shoulder surgery or those with a history of multiple shoulder surgeries
* Concomitant severe glenohumeral arthritis or adhesive capsulitis
* Patients with a worker's compensation claim
* Patients diagnosed with psychological disorders
* Patients with a history of alcohol or drug abuse -Patients on preoperative narcotic therapy -

Min Age: 15 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All athletes undergoing arthroscopic capsulolabral repair surgery will be eligible for participation
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2018-05-14 (Actual); Primary Completion 2021-05 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Successful completion of the return to play checklist | 1 year post-surgery
  This outcome measure will count the number of patients who meet all the criteria in the return to play checklist prior to returning to their sport

CONTACTS AND LOCATIONS:
Locations (1):
- Rothman Orthopaedics at Egg Harbor Township, Egg Harbor, New Jersey, United States